CLINICAL TRIAL: NCT07014046
Title: Simple Bed Exercises for Reducing Postoperative Ileus in Colorectal Surgical Patients, a Randomized Controlled Trial
Brief Title: Simple Bed Exercises for Reducing Postoperative Ileus in Colorectal Surgical Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Shuk-Ting, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIRB-2024-115-1
Record Dates: First submitted 2025-05-27; First posted 2025-06-10 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Ileus
Keywords: postoperative ileus; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simple bed exercises arm (Experimental): The participants will be asked to perform exercise by lying flat on bed in supine position with their eyes look towards to the ceiling of the ward and start focusing on deep breathing exercises with slow inhalations and exhalations. These exercises aim to achieve regular pattern of abdominal muscles and improve the coordination between breathing, abdominal muscle contractions and colonic propulsions. After one-minute deep-breathing exercises, intervention group participants will be asked to pull both knees towards chest in return and turning body from one side to another while lying on bed.
  Interventions: Other: Simple bed exercises
- control arm (No Intervention): usual care

INTERVENTIONS:
Other: Simple bed exercises — The participants will be asked to perform exercise by lying flat on bed in supine position with their eyes look towards to the ceiling of the ward and start focusing on deep breathing exercises with slow inhalations and exhalations. These exercises aim to achieve regular pattern of abdominal muscles and improve the coordination between breathing, abdominal muscle contractions and colonic propulsions. After one-minute deep-breathing exercises, intervention group participants will be asked to pull both knees towards chest in return and turning body from one side to another while lying on bed.
  Arms: Simple bed exercises arm

SUMMARY:
The purpose of this study is to examine the effect of simple bed exercises for reducing postoperative ileus among colorectal surgical patients who have completed colorectal surgery and are experiencing postoperative ileus. The research team will recruit participants in list of elective colorectal surgeries from the Department of Surgery in the United Christian Hospital. The potential participants will first be assessed for eligibility by completing a simple screening assessment, which may take 10 minutes at facilities within the United Christian Hospital. If the patients meet the inclusion criteria, they will continue to take part in the study.

The participants will be assigned randomly (1:1) to either Group 1 or Group 2 via computer randomization. Participants of Group 1 will receive education for simple bed exercises after colorectal surgery. Participants will be asked to have simple bed exercises for 15 minutes, three times a day starting from postoperative day one, until passing the first stool after surgery. All sessions will be conducted by surgical nurse in the United Christian Hospital. Surgical nurses will educate simple bed exercises with exercise video. Participants will be instructed to practise the simple bed exercises 3 times per day for 15 minutes each time at before breakfast, before lunch and before dinner, on top of the standard usual care. Participants in Group 2 will be placed under control group to receive standard usual care.

All participants are required to record defecation, flatus and tolerance of oral intake starting from postoperative day one. Records will take place at 3-time points for both groups: at breakfast, at lunch and at dinner time. Each time participants must complete one set of record on the logbook provided by nurses. If necessary, clinical records including medical history and follow-up appointment time will be retrieved from electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged >/=18 years,
* patients who are diagnosed with colorectal problems that require elective colorectal surgical intervention either anastomosis or stoma, either open or laparoscopic, and the use of any type of postoperative analgesic,
* orientate to have informed consent and who have signed informed consent.

Exclusion Criteria:

* Patients who are not in the list of elective colorectal surgeries
* Patients who require intraoperative and long postoperative intensive care >1 day,
* with a history of mental disorder or confusion,
* patients with any active limitation which affects adherence to the study procedures like severe dementia and physical limitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to first defecation | after surgery until first defecation (up to 7 days after operation)
  Time to first defecation is defined as the interval between the end of the operation and the first observed passage of stool from rectum/ stoma. It will be observed via the stoma bag if defecation occur or by asking the patients or by reviewing the input and output chart when changing diapers for patients. All this observation will be done by nurses. Time to first defecation is expected to be shorter in intervention group if the intervention is effective for solving postoperative ileus as bowel movement resume faster. Time to first defecation is reliable as no defecation implied postoperative ileus.

SECONDARY OUTCOMES:
time to first flatus | after surgery until first flatus (up to 7 days after operation).
  Time to first flatus is defined as the interval between the end of the operation and the first passage of flatus via rectum reported by patients or in stoma bag observed by nurses. The intervention is expected to be effective if it takes a shorter time to first flatus for intervention group than that of the control group.
tolerance to oral diet | after surgery until tolerance of oral diet without any nausea and vomiting (up to 15 days after operation).
  Time to tolerate oral diet is defined as tolerance of oral diet for at least 24 hours without any nausea and vomiting. Patients who do not tolerate oral diet will have symptoms of nausea and vomiting as postoperative ileus occur. Nasogastric tubes will be inserted to prevent aspiration and total parenteral nutrition will be applied and keep patient for sips of water or nil by mouth except medications to allow time for solving postoperative ileus in hospital stays.

CONTACTS AND LOCATIONS:
Locations (1):
- United Christian Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided